CLINICAL TRIAL: NCT05474716
Title: The Effect of Topical Brimonidine on the Hemodynamics of the Optic Nerve Head and Retinochoroidal Circulation in Patients of Primary Open Angle Glaucoma Using Optical Coherence Tomography Angiography
Brief Title: The Effect of Topical Brimonidine on the Ocular Hemodynamics in Patients of POAG Using OCTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Ameen Ismail, Research assistant of ophthalmology, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M 488
Record Dates: First submitted 2022-01-30; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Blood Flow; Optical Coherence Tomography Angiography
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Brimonidine Tartrate; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: A longitudinal, prospective, interventional, uncontrolled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Brimonidine 0.2% bid ophthalmic solution (Experimental): Topical Brimonidine tartrate 0.2% ophthalmic solution used twice daily. It is a selective alpha 2 adrenergic agonist that is used as an ocular hypotensive in glaucoma and ocular hypertension patients and has proposed neuroprotective effect.
  Interventions: Drug: Brimonidine tartrate 0.2% ophthalmic solution

INTERVENTIONS:
Drug: Brimonidine tartrate 0.2% ophthalmic solution — Topical Brimonidine tartrate 0.2% bid ophthalmic solution. A selective alpha 2 adrenergic agonist with ocular hypotensive and neuroprotective properties used in glaucoma and ocular hypertension.

SUMMARY:
Topical Brimonidine is a well-established topical antigalucoma, ocular hypotensive therapeutic that has been in use since 1996. Brimonidine stands out among other topical ocular hypotensives in that it has a neuroprotective effect that is independent of IOP reduction. This has been demonstrated in multiple animal and human controlled studies both in vivo and in vitro. The mechanisms proposed so far to account for this neuroprotection focus mainly on molecular level antiapoptotic effects and modulation of some excitatory stimuli like glutamate. In this study we try to test the hypothesis that a positive hemodynamic profile of Brimonidine on ocular blood flow may be responsible at least in part for its unique neuroprotective effects.

DETAILED DESCRIPTION:
* Study Design: A prospective, longitudinal, interventional, uncontrolled study
* Participants: primary open angle glaucoma patients recruited during the period of study from the fayoum university hospital ophthalmic outpatient clinic.
* Methods:

Primary open angle glaucoma patients that are Brimonidine naiive and at the same time either medication naiive or have been on a fixed antiglaucoma medication for at least a month prior will be commenced on Brimonidine 0.2% bid with prior baseline imaging by OCT angiography (Optovue) of macula 6*6 mm and ONH 4.5*4.5 mm. After commencing Brimonidine patients will be followed up by OCT angiography at three visits assigned for 1,2,3 months after commencing Brimonidine. Every time the patient is imaged by OCT, imaging is done twice, once in a seated position at presentation and another- also in a seated position-, but after a protocol of right recumbency for 30 minutes in order to produce a postural position change as a vascular stress test to assess autoregulatory capacity of ocular and systemic circulation.

At each visit, IOP and arterial blood pressure are measured both in the seated position and after the 30-minute recumbency protocol in order to mathematically calculate the mean ocular perfusion pressure that will be correlated with OCT angiography data including vascular density, as well as indirect parameters of blood flow.

Data will be statistically analysed using the SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma patients.
* Brimonidine naiive.
* Medication naiive or on a fixed antiglaucoma medication for at least a month prior to commencing Brimonidine.

Exclusion Criteria:

* Glaucomas other than primary open angle glaucoma.
* Other comorbid diseses both ocular and systemic that might confound the density and flow measurements ( hypertension, diabetes, vasculitis, MacTel, Uveitis)
* Comorbid diseases that constitute relative or absolute contraindication to Brimonidine ( pregnancy, lactation, bronchial asthma, cardiovascular diseases)
* Prior use of Brimonidine.
* A change in the glaucoma medication regimen within Less than one month at time of presentation.
* Allergy to Brimonidine or related compounds.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in macular and peripapillary vascular densities | At baseline before Brimonidine and 1,2,3 months thereafter.
  The vascular density measured by optical coherence tomography angiography represents the percentage area of flow-positive regions compared to the whole imaged area. Measured densities include (superficial and deep vascular densities) both of the macular area as well as radial peripapillary capillary density of the parapapillary area.
Change in macular and peripapillary flow indices | At baseline before Brimonidine and 1,2,3 months thereafter.
  An arbitrary flow index will be indirectly calculated using the density data of optical coherence tomography angiography, intraocular pressure and arterial blood pressure measurements.

SECONDARY OUTCOMES:
Change in intraocular pressure | At baseline before Brimonidine and 1,2,3 months thereafter.
  Comparing intraocular pressure measurements at baseline with those on subsequent visits.
Change in vascular autoregulatory capacity | At baseline before Brimonidine and 1,2,3 months thereafter.
  Assessing both systemic as well as ocular vascular autoregulatory capacity making use of the 30-minute recumbency protocol as a vascular stress test.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospitals, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No